CLINICAL TRIAL: NCT07405229
Title: Investigation of RIsk Factors in Out-of-hospital-cardiac-arrest Patients, and MEdical Treatment in Idiopathic Ventricular Fibrillation Patients
Brief Title: MEdical Treatment in Idiopathic Ventricular Fibrillation Patients
Acronym: RIME-IVF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bo Gregers Winkel (Other)
Collaborators: The Novo Nordisk Foundation (Unknown); Per Henriksen Foundation (Unknown); Danish Heart Foundation (Other); RH research funds (Unknown)
Responsible Party: Sponsor-Investigator, Bo Gregers Winkel, Chief Physician, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-518057-41-00; 2018-001683-37 (EudraCT Number); H-18017757 (Other: The Regional Research Ethics Committees Denmark)
Record Dates: First submitted 2026-01-26; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Ventricular Fibrillation; Cardiac Arrest, Out-Of-Hospital
Keywords: Idiopathic Ventricular Fibrillation; IVF; cardiac arrest; beta-blocker; treatment; ventricular tachyarrhythmias; Risk markers; quality of life; QoL
MeSH Terms: conditions — Paroxysmal ventricular fibrillation; Out-of-Hospital Cardiac Arrest; Heart Arrest; Tachycardia, Ventricular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beta-blocker (Active Comparator)
  Interventions: Drug: Beta-blocker treatment group
- No medication (No Intervention): Standard care

INTERVENTIONS:
Drug: Beta-blocker treatment group — The betablocker given to the patient will be prioritized: 1) A non-selective betablocker: Propranolol Retard 80 mg daily or Nadolol 40 mg daily OR 2) A selective betablocker: Atenolol 25 mg daily, Bisoprolol 2.5 mg daily or Metoprolol 50 mg.
  Arms: Beta-blocker

SUMMARY:
A person who has experienced a cardiac arrest with no apparent cause is at risk of having recurrent cardiac arrest. Hence an implantable cardioverter-defibrillator (ICD) is recommended on empirical grounds. Today, there is no uniform way of approaching prevention of recurrence in idiopathic ventricular fibrillation (IVF) patients, beside ICD implantation. Better reatment and risk stratification tools are needed Medical treatment in these patients has never been assessed systematically, but at least some patients with no apparent diagnosis are on betablocker treatment. It is not known if low-doselow dose betablocker treatment is beneficial in these patients.

This study investigates the effect of betablocker treatment to reduce arrhythmic burden in IVF patients.

No predictors for appropriate ICD therapy have been identified in patients with IVF. It is also explored if toxicological and/or genetic profiles, together with in depth machine learning simulation data on repolarization patterns from IVF-ECGs compared to controls, can be used as risk stratification tools.

Lastly, QOL in IVF patients and the impact of beta blocker treatment will be investigated.

ELIGIBILITY:
Inclusion Criteria:

Resuscitated OHCA patients admitted to one of the participating hospitals.

1. Age ≥18 years
2. Suspected cardiac cause of cardiac arrest

Exclusion Criteria:

OHCA patients

1. With Ischemic heart disease.
2. Obvious non-cardiac cause of cardiac arrest
3. Congenital heart disease
4. Do not speak or understand Danish
5. Foreigners -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
First appropriate therapy by ICD or 3 years after discharge | 3 years
  Primary outcome will be either first appropriate therapy by ICD (anti tachycardia pacing or DC conversion), or aborted shock or non-sustained ventricualr fibrillation detected by the ICD, where the treating physician opts for a change in medication, or no therapy from the ICD 3 years after randomization, whichever comes first.

SECONDARY OUTCOMES:
Quality of Life at 3 months | 3 months
  Quality of life will be assessed by trained nurses. Focus will be on betablocker therapy and overall cognitive abilities after cardiac arrest. Patients will be assessed using the SF-36 (v1) quality of life tool. The patients will be assessed 3 months after discharge.
Quality of Life at 1 year | 1 year
  Quality of life will be assessed by trained nurses. Focus will be on betablocker therapy and overall cognitive abilities after cardiac arrest. Patients will be assessed using the SF-36 (v1) quality of life tool. The patients will be assessed 3 1 year after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Bo G Winkel, MD, Principal Investigator — The Heart Center, Rigshospitalet
Locations (2):
- Denmark (2):
  - The Heart Center, Rigshospitalet, Copenhagen, Dr.
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No
GDPR